CLINICAL TRIAL: NCT05952024
Title: A Prospective, Open-Label, Single-Arm, Phase II Study of Acalabrutinib and Rituximab in Untreated Elderly and/or Frail Patients With Diffuse Large B-Cell Lymphoma (ACRUE)
Brief Title: Study of Acalabrutinib and Rituximab in Untreated Elderly and/or Frail Patients With DLBCL
Acronym: ACRUE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8227C00002
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Chemoimmunotherapy treatments; Treatment-naïve elderly patients
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — acalabrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib and Rituximab (Experimental): Patients will receive Dose A of acalabrutinib orally in X dosing schedule beginning on Cycle 1 Day 1 for a maximum of 28 cycles or until 2014 Lugano Classification for Non-Hodgkin's Lymphoma (NHL)-defined disease progression or another discontinuation criterion is met. Patients will also receive an intravenous (IV) infusion of Dose B rituximab on Cycle 1 Day 15 and Dose C of rituximab as an subcutaneous (SC) injection on Day 1 of Cycle 2 through Cycle 8.
  Interventions: Drug: Acalabrutinib; Biological: Rituximab

INTERVENTIONS:
Drug: Acalabrutinib — Patients will receive acalabrutinib orally with dosing schedule of X.
  Other Names: CALQUENCE®
Biological: Rituximab — Patients will receive rituximab via IV infusion on Cycle 1 Day 15 and via SC injection on Day 1 of Cycle 2 through Cycle 8.

SUMMARY:
The study will measure the safety, tolerability, and efficacy with acalabrutinib in combination with rituximab in treatment-naïve elderly and/or frail patients with diffuse large B-cell lymphoma (DLBCL), who are otherwise unsuitable for standard front line chemoimmunotherapy treatments.

DETAILED DESCRIPTION:
Treatment-naïve elderly and/or frail patients with DLBCL will be treated with acalabrutinib in combination with rituximab in a single arm.

Study details include the following:

* The study duration will be up to 108 weeks for each patient, including up to 28 days for screening and 104 weeks of treatment and follow-up.
* The treatment duration will be up to 8 cycles for rituximab and 28 cycles for acalabrutinib both beginning at cycle 1.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 80 years of age at the time of screening, or
* ≥ 65 to 79 years of age at the time of screening and considered ineligible for chemoimmunotherapy
* Histologically documented DLBCL
* No prior treatment for DLBCL
* Stage II, III, or IV disease by the Ann Arbor Classification .
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2 with no deterioration over the previous 2 weeks prior to baseline or day of the first dosing except when due to underlying lymphoma.
* At least 1 lesion that can be accurately measured at baseline as ≥ 10 mm in the longest diameter with computed tomography or magnetic resonance imaging and is suitable for accurate repeated measurements.
* Adequate organ and marrow function independent of growth factor or transfusion support within 1 week of Screening.

Exclusion Criteria:

* Any evidence of diseases (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension, renal transplant, and active bleeding diseases), that would make the study undesirable for the patient or that would impact compliance with the protocol.
* History of prior or current malignancy, that would affect compliance with the protocol or interpretation of the results.
* Serologic status reflecting active hepatitis B or C infection.
* Serological positivity or known infection with HIV.
* Active central nervous system involvement by lymphoma, leptomeningeal disease, or spinal cord compression.
* Any comorbidity or organ system impairment rated with a single Cumulative Illness Rating Scale-Geriatric score (CIRS-G) of 4 or a total CIRS-G score of > 17.
* History of or ongoing confirmed Progressive Multifocal Leukoencephalopathy.
* Known active significant infection.
* History of stroke or intracranial haemorrhage within 6 months before the first dose of study drug.
* History of bleeding diathesis (eg, haemophilia, von Willebrand disease).
* Major surgical procedure within 30 days of first dose of study intervention or anticipated major surgery during the study timeframe.
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists.
* Received a live virus vaccination within 28 days of the first dose of study drug.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2027-08-24 (Estimated); Study Completion 2027-08-24 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with Grade 3 to 4 treatment emergent adverse events (TEAEs) | Cycle 1 Day 1 (Cycles 1 to 8 is 21 days and Cycles 9 to 28 is 28 days) through End of treatment EoT [30 days of discontinuation] (Up to 3.5 Years)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Cycle 1 Day 1 (Cycles 1 to 8 is 21 days and Cycles 9 to 28 is 28 days) Until disease progression or last evaluable assessment in the absence of progression (Up to 3.5 Years)
Progression free survival (PFS) | Cycle 1 Day 1 (Cycles 1 to 8 is 21 days and Cycles 9 to 28 is 28 days) Until disease progression or last evaluable assessment in the absence of progression (Up to 3.5 Years)
Event-Free Survival (EFS) | Cycle 1 Day 1 (Cycles 1 to 8 is 21 days and Cycles 9 to 28 is 28 days) Until disease progression or last evaluable assessment in the absence of progression (Up to 3.5 Years)
Overall survival (OS) | Cycle 1 Day 1 (Cycles 1 to 8 is 21 days and Cycles 9 to 28 is 28 days) Until Post-treatment follow-up (Up to 3.5 Years)
Duration of response (DoR) | Cycle 1 Day 1 (Cycles 1 to 8 is 21 days and Cycles 9 to 28 is 28 days) Until disease progression or last evaluable assessment in the absence of progression (Up to 3.5 Years)
Change from baseline in Timed Up and Go test (TUG) | Cycle 1 Day 1 (Cycles 1 to 8 is 21 days and Cycles 9 to 28 is 28 days) Until Post-treatment follow-up (Up to 3.5 Years)
Number of patients with adverse events | Screening (up to 28 days before day 1) Until Post-treatment follow-up (Up to 3.5 Years)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (10):
  - Research Site, La Jolla, California
  - Research Site, Orange, California
  - Research Site, Jacksonville, Florida
  - Research Site, Waukee, Iowa
  - Research Site, Baltimore, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Lubbock, Texas
  - Research Site, Olympia, Washington
  - Research Site, Tacoma, Washington
- Brazil (16):
  - Research Site, São Paulo, Barretos
  - Research Site, Minas Gerais, Belo Horizonte
  - Research Site, Distrito Federal, Brasilia
  - Research Site, São Paulo, Campinas
  - Research Site, Paranã, Curitiba
  - Research Site, Santa Catarina, Florianopolis
  - Research Site, Goiás, Goiania
  - Research Site, Rio Grande Do Norte, Natal
  - Research Site, Rio Grande, Porto Alegre
  - Research Site, Pernambuco, Recife
  - Research Site, São Paulo, Ribeirao Prieto
  - Research Site, São Paulo, Sao Jose Do Rio Preto
  - Research Site, Maranhão, Sao Luis
  - Research Site, São Paulo, Sorocaba
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Research Site, San Juan, Puerto Rico
- South Korea (13):
  - Research Site, Busanjin-gu, Busan
  - Research Site, Seo-gu, Busan
  - Research Site, Dalseo-gu, Daegu
  - Research Site, Namdong-gu, Incheon
  - Research Site, Jeollabuk-do, Jeonju-si
  - Research Site, Gyeongsangnam-do, Jinju-si
  - Research Site, Gangnam-gu, Seoul
  - Research Site, Seocho-gu, Seoul
  - Research Site, Seodaemun-gu, Seoul
  - Research Site, Songpa-gu, Seoul
  - Research Site, Yangch’ŏn-gu, Seoul
  - Research Site, Gyeonggi-do, Suwon-si
  - Research Site, Dong-gu, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/